CLINICAL TRIAL: NCT02432768
Title: The Effect of Triheptanoin in Adults With McArdle Disease (Glycogen Storage Disease Type V)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other); University of Texas Southwestern Medical Center (Other); Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Principal Investigator, Karen Lindhardt Madsen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-8-2014-006; 2014-003644-12 (EudraCT Number)
Record Dates: First submitted 2014-11-04; First posted 2015-05-04 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Glycogen Storage Disease Type V
Keywords: Anaplerotic diet; McArdle Disease; Glycogen Storage Disease; Triheptanoin
MeSH Terms: conditions — Glycogen Storage Disease Type V; Glycogen Storage Disease | interventions — triheptanoin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triheptanoin (Active Comparator): 14 days on Triheptanoin treatment including a 7 days titration period and a 7 days full dose treatment of 1mL/kg/day.
  Interventions: Drug: Triheptanoin
- Placebo oil (Placebo Comparator): 14 days of diet on a placebo oil including 7 days titration period and 7 days full dose treatment of 1mL/kg/day.
  Interventions: Other: Placebo oil

INTERVENTIONS:
Drug: Triheptanoin — Anaplerotic dietary oil
  Other Names: UX007
  Arms: Triheptanoin
Other: Placebo oil — Safflower oil
  Other Names: UX007 Placebo Oral Liquid
  Arms: Placebo oil

SUMMARY:
Background: Patients with the sugar metabolism disorder, Glycogen Storage Disease Type V, have insufficient breakdown of sugar stored as, glycogen, within the cells. The investigators know from previous studies with McArdle patients, that they not only have a reduced sugar metabolism, both also have problems in increasing their fat metabolism during exercise to fully compensate for the energy deficiency.

Studies on Triheptanoin diet used in patients with other metabolic diseases have shown that Triheptanoin can increase metabolism of both fat and sugar. In these patients, Triheptanoin has had a positive effect on the physical performance and has reduces the level of symptoms experienced by patients.

Aim: To investigate the effect of treatment with the dietary oil, Triheptanoin, in patients with McArdle disease on exercise capacity.

Methods: 20-30 adult patients will be recruited through Rigshospitalet in Copenhagen, Denmark, Hopital Pitié-Sapêtrière in Paris, France and through The University of Texas Southwestern Medical Center in Dallas, Texas.

1. Pre-experimental testing (1 day):

   Baseline blood samples are collected to obtain baseline values of safety parameters: Plasma-acylcarnitines, free fatty acids and creatine kinase.

   Subjects perform a max-test to determine their VO2max
2. Treatment period #1 (2 weeks):

   Subjects follow a diet consuming a dietary treatment oil. Neither patients nor members of the study group know who receive which type of oil.
3. Washout period (1 week):

   Subjects receive no treatment
4. Treatment period #2 (2 weeks):

Subjects who received Triheptanoin oil in the first treatment period, now receive placebo oil and vice versa.

Assessments: Before and after each treatment periods, subjects perform a 30-minutes exercise test on a cycle ergometer, comprising of 20-22 minutes of constant load exercise and 6-8 minutes increasing load to peak. Subjects will complete a Fatigue Severity Scale questionnaire and metabolic products will be measured in blood and urine.

DETAILED DESCRIPTION:
BACKGROUND

This project will investigate the treatment potential of the drug Triheptanoin in patients with the inborn defect in glycogen metabolism, McArdle Disease. There is currently no treatment available for this group of patients. The condition leads to intolerance to physical exercise with a risk of developing severe cramps and contractures followed by muscle damage and acute kidney failure. Also one third of the patients develop progressive muscle weakness and wasting.

The McArdle patients have an inherited defect in the enzyme, myofosforylase, an important link in the glycogenolysis within skeletal muscle. As a consequence, the patients lack substrates for glycolysis to fuel muscle work (1). The investigators have previously shown that patients with McArdle disease are unable to increase fat metabolism enough to compensate for the energy insufficiency that occurs in these patients in response to exercise (2).

A key limitation to exercise in McArdle disease is the reduced production of pyruvate, causing depletion of intermediates in the Citric Acid Cycle (CAC). Triheptanoin is a triglyceride of glycerol and three 7-carbon fatty acid chains (heptanoate). The breakdown of odd-number carbon fatty acids, such as heptanoate, generates CAC-intermediates. Triheptanoin can therefore potentially boost the flux through the CAC and increase the ATP and energy generation in the cells.

In other patients with inborn errors of metabolism, treatment with daily Triheptanoin supplement can increase metabolism of both fat and glucose. Triheptanoin treatment has reduced the symptom frequency and increased exercise tolerance and physical performance in these patients (3,4).

The aim of this study is to investigate the effect of Triheptanoin on exercise performance and tolerance and frequency of symptoms in patients with McArdle disease.

METHODS

The study will be designed as a double blinded placebo controlled cross-over study. During a 5 week trial period each study patient will go through a 2 week treatment period, a 1 week wash-out period without treatment followed by another 2 week treatment period. In one treatment period, the patient takes a daily dietary oil supplement containing Triheptanoin and in the other period, the oil contains regular safflower oil (placebo). Both Triheptanoin and placebo oil is manufactured, packed and handed out by the manufacturer, Ultragenyx Pharmaceuticals Inc. in a way that neither patients, nor the investigators will know in which period, which treatment is given to which patient.

Assessments:

The patients will meet at the laboratory for assessments on 5 occasions:

* Screening visit: Patients perform a peak exercise test on a cycle ergometer wearing a mask that can measure oxygen and carbon dioxide exchange rates. Patients exercise with increasing workload until exhaustion to find their maximal oxidative capacity and maximal workload
* Test days 1-4: On one test day before and one after each treatment period, the patients perform a 30-minutes exercise test on a cycle ergometer working at a constant moderate intensity for 20-22 minutes followed by a 6-8 minutes stepwise increase to peak workload. Blood samples will be taken before, during and after exercise to measure concentrations of metabolic products. Patients report their current feeling of fatigue in a Fatigue Severity Scale (FSS-questionnaire)

Subjects:

A total number of 21-28 patients will be included in the study across three trial sites. From the Danish cohort of McArdle Patients; 5-8 patients will be included and from the French cohort; 8-10 patients will be included and from the 8-10 American patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Genetically and/or biochemically verified diagnosis of McArdle disease
* Body Mass Index of 18-32
* Capacity to consent

Exclusion Criteria:

* Significant cardiac and pulmonary disease
* Pregnancy
* Treatment with beta-blockers
* Inability to perform cycling exercise
* Any other significant disorder that may confound the interpretation of the findings

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in heart rate during constant load cycling exercise (HRconst) with Triheptanoin vs. placebo treatment | Day 14 and day 28
  Subject heart rate will be measured during 20 minutes exercise test performed on a cycle ergometer at a workload corresponding to approximately 60% of maximal oxidative capacity (VO2max).

SECONDARY OUTCOMES:
Change in maximal oxidative capacity (VO2max) with Triheptanoin vs. placebo treatment | Day 14 and day 28
  The maximal oxidative capacity measured at peak workload after a 6 minutes ramp test performed on a cycle ergometer after 20 minutes constant load cycling.
Change in self-rated severity of fatigue symptoms with Triheptanoin vs. placebo treatment | Day 14 and day 28
  Total score on a Fatigue Severity Scale (FSS)
Change in urine concentrations of organic acids with Triheptanoin vs. placebo treatment | Day 14 and day 28
  Urine concentrations of: 3OH-propionate, heptanoate, methylmalonate, pimelate methylcitrate
Change in maximal workload capacity (Wmax) with Triheptanoin vs. placebo treatment | Day 14 and day 28
  The maximal workload capacity (Wmax) is measured at peak workload after a 6 minutes ramp test performed on a cycle ergometer after 20 minutes constant load cycling.
Change in plasma concentrations of metabolites, citric acid cycle (CAC) intermediates with Triheptanoin vs. placebo treatment | Day 14 and day 28
  Plasma concentrations of metabolites and citric acid cycle (CAC) intermediates: Lactate, ammonia, glucose, Free Fatty Acids (FFA), acyl-carnitines and malate (a CAC intermediate).

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Madsen, MD, Principal Investigator — Neuromuscular Research Unit, Rigshospitalet
Locations (1):
- Copenhagen Neuromuscular Center, 3342, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Mommaerts WF, Illingworth B, Pearson CM, Guillory RJ, Seraydarian K. A FUNCTIONAL DISORDER OF MUSCLE ASSOCIATED WITH THE ABSENCE OF PHOSPHORYLASE. Proc Natl Acad Sci U S A. 1959 Jun;45(6):791-7. doi: 10.1073/pnas.45.6.791. No abstract available. PMID 16590445
- [Background] Orngreen MC, Jeppesen TD, Andersen ST, Taivassalo T, Hauerslev S, Preisler N, Haller RG, van Hall G, Vissing J. Fat metabolism during exercise in patients with McArdle disease. Neurology. 2009 Feb 24;72(8):718-24. doi: 10.1212/01.wnl.0000343002.74480.e4. PMID 19237700
- [Background] Roe CR, Sweetman L, Roe DS, David F, Brunengraber H. Treatment of cardiomyopathy and rhabdomyolysis in long-chain fat oxidation disorders using an anaplerotic odd-chain triglyceride. J Clin Invest. 2002 Jul;110(2):259-69. doi: 10.1172/JCI15311. PMID 12122118
- [Background] Roe CR, Yang BZ, Brunengraber H, Roe DS, Wallace M, Garritson BK. Carnitine palmitoyltransferase II deficiency: successful anaplerotic diet therapy. Neurology. 2008 Jul 22;71(4):260-4. doi: 10.1212/01.wnl.0000318283.42961.e9. PMID 18645163
- [Background] Stojkovic T, Vissing J, Petit F, Piraud M, Orngreen MC, Andersen G, Claeys KG, Wary C, Hogrel JY, Laforet P. Muscle glycogenosis due to phosphoglucomutase 1 deficiency. N Engl J Med. 2009 Jul 23;361(4):425-7. doi: 10.1056/NEJMc0901158. No abstract available. PMID 19625727